CLINICAL TRIAL: NCT06678906
Title: Physical Inactivity and Sedentary Behavior: Screening and Intervention in Ambulatory Primary Care
Acronym: IPSEDI
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Grenoble (Other)
Collaborators: Clinical Investigation Center - University Hospital Grenoble (Unknown); Department of Physiotherapy - Grenoble Alpes University - TIMC LAboratory (UMR-UGA-CNRS-5525) (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Supportive Care
Other Study IDs: 38RC23.031
Record Dates: First submitted 2024-10-14; First posted 2024-11-07 (Actual); Last update posted 2025-02-10 (Actual); Status verified 2025-02

CONDITIONS: Primary Care
Keywords: Physical inactivity; Sedendary behavior; Innovative personalized support by physiotherapist; Ambulatory primary care; Healthcare pathway
MeSH Terms: conditions — Sedentary Behavior

STUDY DESIGN:
Intervention Model Description: Cluster randomization will be conducted according to the "stepped wedge" design.
Masking Description: As a result, all centers will include patients both before (control period) and after the implementation of the intervention (experimental period). The timing of the intervention implementation (training period) for each center will be randomized among 4 training periods distributed throughout the study, with two centers per training period
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control arm (No Intervention): Control group will receive standard information about physical activity and sedentary lifestyle.
- Intervention arm (Experimental): All patients in the intervention group will benefit from the standard information phase on physical activity and sedentary behavior, as well as personalized support for behavior change in the form of a serious game and remote coaching.
  Interventions: Behavioral: Intervention arm

INTERVENTIONS:
Behavioral: Intervention arm — All patients in the intervention group will benefit from the standard information phase on physical activity and sedentary behavior, as well as personalized support for behavior change in the form of a serious game and remote coaching.
  Arms: Intervention arm

SUMMARY:
Physical inactivity and sedentary behaviors are among the leading modifiable risk factors for chronic diseases. In France, despite the national Sport Health strategy, awareness campaigns physical inactivity and sedentary behavior worsened between 2005 and 2015. Primary healthcare professionals, including general practitioners and physiotherapists already involved in tertiary prevention, can act for primary and secondary prevention.

DETAILED DESCRIPTION:
In this study, we hypothesize that an innovative care pathway based on opportunistic screening by general practitioners to assess levels of physical activity and sedentary behavior, and an individualized intervention by a physiotherapist effectively supports behavioral changes towards increased physical activity and reduced sedentary behavior at 6 months in inactive adults without chronic conditions.

This multicenter study, employing an innovative stepped-wedge cluster methodology, will enable healthcare professionals from all included multidisciplinary health centers to enhance their skills in supporting health behavior changes.

For all patients, participation in the study should lead to an increased awareness of the risks associated with physical inactivity and sedentary behaviors.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients
* Not benefiting from Long-Term Illness coverage
* Followed in primary outpatient care by one of the participating centers
* Patients identified as "inactive" by the ONAPS-PAQ questionnaire during an appointment with a general practitioner in the partner Multi-Professional Health Centers, whether sedentary or not
* Patient having signed informed consent to participate in the study
* Patients who understand and speak French
* Persons affiliated with a social security scheme or beneficiaries of a similar scheme
* Patients classified as "inactive" (< 600 MET.min/week) after 7-day actimetry analysis

Exclusion Criteria:

* Patient receiving follow-up for another reason with physiotherapists participating in the protocol
* Persons referred to in articles L1121-5 to L1121-8 of the Public Health Code
* Patient participating in another interventional research study with an exclusion period still ongoing at pre-inclusion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2025-05 (Estimated); Primary Completion 2027-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Evaluate the 6-month effectiveness of an individualized intervention by a physiotherapist, on physical activity and sedentary behavior in adult patients without chronic diseases | 6 months
  1. Proportion of patients changing to a higher physical activity category, measured by actimetry, between inclusion and M6, defined as: from inactive to moderately active or very active
  2. Proportion of patients changing to a lower sedentary behavior category, measured by actimetry, between inclusion and M6, defined as: from high sedentary behavior to moderate sedentary behavior or non-sedentary and from moderate sedentary behavior to non-sedentary

SECONDARY OUTCOMES:
Describe the evolution of patients' physical activity and sedentary behavior levels at 6 months (for behavior change) and 12 months (for behavior maintenance). | 12 months
  ONAPS-PAQ questionnaire score
Quantify the evolution of patients' physical activity and sedentary behavior levels at 6 months (for behavior change) and 12 months (for behavior maintenance). | 12 months
  7-day accelerometry measurement
Explore the relationship between patient characteristics and changes (at 6 months) and maintenance (at 12 months) of physical activityand sedentary behavior levels. | 12 months
  Degree of correlation between the socio-demographic categories (age, sex, socio-economic category, environment and place of residence, type and work hours) and 7-day accelerometry measurement
Describe the quality of motivation initially (Month 0), at 6 months, and at 12 months. | 12 monts
  MAPS questionnaire score
Describe the satisfaction of basic psychological needs at 6 months, and at 12 months. | 12 monts
  Basic Psychological Needs Scale score
Describe the self-efficacy perceived competence scale for engaging in a personalized physical activity program at 6 months and at 12 months. | 12 monts
  Score obtained at perceived competence scale for engaging in a personalized physical activity program
Describe the perceived level of vitality and energy initially (M0), at 6 months, and at 12 months. | 12 monts
  Score obtained at perceived vitality and energy scale
Describe the self-esteem initially (M0), at 6 months, and at 12 months. | 12 monts
  Score obtained at the self-esteem scale
Describe at M6 and M12 the strategies, barriers, and facilitators to patients' behavior change. | 12 months
  Extraction of coaching verbatims coupled with a qualitative survey using semi-structured interviews on a sample of volunteer patients who may or may not have benefited from the intervention at 6 months and 12 months.
Study the relationship between ONAPS-PAQ results and 7-day actimetry in this population category (inactive and/or sedentary). | 12 months
  Degree of correlation between categorizations obtained by energy expenditure from accelerometry and the ONAPS-PAQ questionnaire
Identify perceived barriers and facilitators to implementation in primary care at 12 months among different stakeholders (general practitioners, physiotherapists, patients). | 12 months
  Score obtained on the scale of level of satisfaction and perception of the project's implementation in primary care by the various players: doctors, physiotherapists and patients.

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas PINSAULT, Professor, Principal Investigator — Physiotherapy department - Grenoble Alpes University
Locations (1):
- Pr Nicolas PINSAULT, Saint-Martin-d'Hères, France

REFERENCES:
- [Derived] Pinsault N, Rey S, Druart L, Guizon AH, Debru R, Roustit M, Pison C. Physical inactivity and sedentary behaviours: screening and intervention in primary care, a prospective, multicentre, cluster-randomised, controlled, stepped-wedge study. BMC Public Health. 2025 Nov 14;25(1):3951. doi: 10.1186/s12889-025-25410-4. PMID 41239336
- See also: Related Info — https://www.anses.fr/fr/system/files/INCA3-ActivitesPhysiques.pdf
- See also: Related Info — https://www.santepubliquefrance.fr/determinants-de-sante/nutrition-et-activite-physique/etude-de-sante-sur-l-environnement-la-biosurveillance-l-activite-physique-et-la-nutrition-esteban-2014-2016.-volet-nutrition.-chapitre-corpulence